CLINICAL TRIAL: NCT04716790
Title: Randomized Clinical Trial to Elucidate the Effects of Low Frequency Ultrasound Debridement (LFU), in Patients With Diabetic Foot Ulcers, Compared to Its Conventional Treatment
Brief Title: Comparison Between the Effect of Ultrasound Debridement and Conventional Treatment in Diabetic Foot Ulcers (DFU).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Yolanda García Álvarez (Unknown); Francisco Javier Álvaro Afonso (Unknown)
Responsible Party: Principal Investigator, Sebastian Flores Escobar, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ultrasound Debridement; 20/738-EC_P (Other: Ethics Committee of the Hospital Clínico San Carlos)
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot; Diabetic Foot Ulcer; Ultrasound Debridement; Ultrasonic Debridement
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: A randomized and controlled parallel clinical trial
Who Masked: Investigator
Masking Description: The clinician who performs the cures, photographs and data collection is different from the clinician who performs the application of ultrasound debridement. Therefore, the evaluator will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ultrasounds once a week (Experimental): Patients will undergo the application of ultrasound therapy with a frequency of once a week.
  Interventions: Procedure: Ultrasound Debridement
- Ultrasounds once every two weeks (Experimental): Patients will undergo the application of ultrasound therapy with a frequency of once every two weeks.
  Interventions: Procedure: Ultrasound Debridement
- Standard of care (Active Comparator): Patients will be treated using the conventional treatment established by the protocol of the Diabetic Foot Unit of the University Podiatry Clinic of Complutense University of Madrid.
  Interventions: Procedure: Conventional Treatment

INTERVENTIONS:
Procedure: Ultrasound Debridement — Ultrasounds debridement is performed using an SONOCA 185 device (Söring GmbH, Germany). The ultrasounds device generates an ultrasound low frequency of 25kHz and is equipped with three instruments with different sonotrode shapes. The choice of sonotrode depends on wound depth. The ultrasounds instrument piezoelectrically transforms the electrical energy delivered from the ultrasound device into mechanical oscillations in the sonotrode tip.
  Arms: Ultrasounds once a week; Ultrasounds once every two weeks
Procedure: Conventional Treatment — Conventional Treatment based on international guidelines for diabetic foot
  Arms: Standard of care

SUMMARY:
The investigators aimed to elucidate the effects of ultrasound debridement on the area and healing of diabetic foot ulcers compared to their conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years old.
* Type 1 or type 2 diabetes mellitus with HbA1c ≤ 10%.
* DFU grades IA, IIA, IB, IIB, IC, IIC, ID, IID, according to the University of Texas Classification.
* DFU grades PEDIS 1-Absence of Infection, PEDIS 2-Mild infection and PEDIS 3-Moderate infection, according to the PEDIS-IDSA Classification.
* Wound size between 1 cm² and 30 cm².
* Evolution time DFU between 1 and 24 months.
* Ankle-brachial index (ABI) ≤0.9 and ankle systolic blood pressure (ASBP) ≥70mmHg, or toe systolic blood pressure (TSBP) ≥50mmHg, ABI>0.9, TSBP ≥50mmHg and toe-brachial index (TBI) ≤0.7

Exclusion Criteria:

* Critical limb ischemia patients with ABI≤0.5 and ASBP<70mmHg or TSBP<50mmHg.
* Clinical suspicion of osteomyelitis.
* Pregnant or lactating women or women of childbearing potential who are not using effective contraception.
* Patients diagnosed with hepatitis or human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-01-18 (Estimated); Study Completion 2023-06-23 (Estimated)

PRIMARY OUTCOMES:
Healing Rate | 12 weeks
  Total epithelialization of the wound.
Healing Time | 12 weeks
  Time from the inclusion of the wound in the study until its total epithelialization.
Wound Size | 12 weeks
  Planimetric measurements of wound size will be made using Visitrak (Smith & Nephew, Hull, UK).

SECONDARY OUTCOMES:
Wound Conditions | 12 weeks
  The wound bed tissue will be evaluated for the presence, quality and consistency of the granulation tissue using a validated wound scoring system, with scores ranging from a minimum of zero points to a maximum of seven points (Wollina Score).
Transcutaneous oxygen pressure (TcPO2) | baseline and week 7
  Two measurements will be made, one at the initial visit and the other at the final visit, and possible variations will be assessed.
Pain intensity | 12 weeks
  It will be assessed using a numerical scale of pain that receives values between zero and ten, understanding zero as the absence of pain and ten as the maximum pain bearable by the patient
Health-related quality of life | baseline and 12 week
  It will be assessed using the SF-36 health-related quality of life questionnaire at the beginning and end of the study. This questionnaire receives values between zero and one hundred so that the higher the score, the better the patient's health status.

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda García Álvarez, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Complutense University, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No